CLINICAL TRIAL: NCT05369832
Title: A Phase 4, Prospective, Open-label Study of Ozanimod to Explore the Safety, Efficacy, Quality of Life, and Biomarker Response in Participants With Moderate to Severe Ulcerative Colitis in Clinical Practice
Brief Title: An Open-label Study of Ozanimod in Moderate to Severe Ulcerative Colitis in Clinical Practice
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM047-029
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis; Ozanimod; RPC-1063; Zeposia®; Inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Advanced therapy-naive (Experimental)
  Interventions: Drug: Ozanimod
- Cohort 2 - Advanced therapy-exposed (Experimental)
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Other Names: Zeposia®; RPC-1063; BMS-986374

SUMMARY:
The purpose of this study is to explore the safety, efficacy, effects on quality of life (QOL), and biomarker response of ozanimod in participants with moderate to severely active ulcerative colitis (UC) in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ulcerative colitis (UC), with signs and symptoms consistent with UC for at least 3 months prior to the first study intervention administration
* Moderate to severely active UC disease activity, defined as a modified Mayo score of 4 through 9, inclusive, with the following minimum subscores:

  i) An SF subscore ≥ 1, AND ii) An RB subscore ≥ 1, AND iii) An ES ≥ 2 (endoscopy performed within 60 days of the first study intervention administration).
* Report of a previous colonoscopy that documents extent of disease

Exclusion Criteria:

* Current or recent (within 3 months of screening) evidence of fulminant colitis, toxic megacolon, or bowel perforation
* Extensive colonic resection or current stoma
* Colonic dysplasia that has not been removed

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (85):
- United States (85):
  - Local Institution - 0048, Dothan, Alabama
  - Local Institution - 0206, Chandler, Arizona
  - Local Institution - 0216, Gilbert, Arizona
  - Local Institution - 0125, Sun City, Arizona
  - Local Institution - 0195, Tucson, Arizona
  - Local Institution - 0045, North Little Rock, Arkansas
  - Local Institution - 0165, Apple Valley, California
  - Local Institution - 0162, Camarillo, California
  - Local Institution - 0014, Lancaster, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Local Institution - 0209, Los Angeles, California
  - Local Institution - 0002, San Diego, California
  - Local Institution - 0208, San Diego, California
  - Local Institution - 0185, San Jose, California
  - Local Institution - 0178, Littleton, Colorado
  - Gastro Florida, Clearwater, Florida
  - Local Institution - 0018, Clearwater, Florida
  - Local Institution - 0050, Homestead, Florida
  - Local Institution - 0026, Lighthouse PT, Florida
  - Local Institution - 0167, Miami, Florida
  - Local Institution - 0049, Miami Lakes, Florida
  - Wellness Clinical Research-Miami Florida, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Local Institution - 0003, Naples, Florida
  - Local Institution - 0058, Orange Park, Florida
  - Local Institution - 0205, Orlando, Florida
  - Local Institution - 0037, Palm Harbor, Florida
  - Local Institution - 0179, Wellington, Florida
  - Local Institution - 0027, Roswell, Georgia
  - Local Institution - 0198, Arlington Heights, Illinois
  - Local Institution - 0051, Chicago, Illinois
  - Local Institution - 0098, Gurnee, Illinois
  - Local Institution - 0192, Kansas City, Kansas
  - Local Institution - 0181, Topeka, Kansas
  - Local Institution - 0183, Louisville, Kentucky
  - Local Institution - 0200, Baton Rouge, Louisiana
  - Local Institution - 0171, Chevy Chase, Maryland
  - Local Institution - 0191, Glen Burnie, Maryland
  - Local Institution - 0199, Boston, Massachusetts
  - Local Institution - 0196, Worcester, Massachusetts
  - Local Institution - 0174, Plymouth, Minnesota
  - Local Institution - 0184, Ocean Springs, Mississippi
  - Local Institution - 0024, Chesterfield, Missouri
  - Local Institution - 0213, Weldon Spring, Missouri
  - Local Institution - 0180, Englewood, New Jersey
  - Local Institution - 0084, Brooklyn, New York
  - Local Institution - 0187, New York, New York
  - Local Institution - 0059, New York, New York
  - NYU Langone Health -Inflammatory Bowel Disease Center, New York, New York
  - Local Institution - 0176, New York, New York
  - Local Institution - 0170, Utica, New York
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Local Institution - 0005, Cincinnati, Ohio
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Local Institution - 0188, Columbus, Ohio
  - Local Institution - 0061, Mentor, Ohio
  - Local Institution - 0060, Providence, Rhode Island
  - Local Institution - 0177, Cordova, Tennessee
  - Local Institution - 0168, Nashville, Tennessee
  - Local Institution - 0038, Bellaire, Texas
  - Novel Research LLC, Bellaire, Texas
  - Local Institution - 0138, Dallas, Texas
  - Local Institution - 0036, Houston, Texas
  - Local Institution - 0163, Houston, Texas
  - Ace Clinical Research Group: Digestive Health Associates, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Local Institution - 0052, Houston, Texas
  - Local Institution - 0129, Katy, Texas
  - Local Institution - 0161, Lubbock, Texas
  - GI Alliance: Mansfield - TDDC, Mansfield, Texas
  - Local Institution - 0039, Mansfield, Texas
  - Local Institution - 0201, San Antonio, Texas
  - Local Institution - 0043, San Antonio, Texas
  - San Antonio Gastroenterology, San Antonio, Texas
  - Local Institution - 0166, San Marcos, Texas
  - Local Institution - 0046, Tyler, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Local Institution - 0091, Webster, Texas
  - Local Institution - 0193, Ogden, Utah
  - Local Institution - 0169, Salt Lake City, Utah
  - Local Institution - 0197, Lynchburg, Virginia
  - Local Institution - 0130, Seattle, Washington
  - Local Institution - 0189, Tacoma, Washington
  - Local Institution - 0017, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 139 participants were enrolled and treated.
Groups:
- Cohort 1: Ozanimod Advanced Therapy Naïve: Advanced therapy naïve participants received ozanimod 0.92 mg daily
- Cohort 2: Ozanimod Advanced Therapy Exposed: Advanced therapy exposed participants received ozanimod 0.92 mg daily
Period: Overall Study
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Started | 99 | 40
Completed | 0 | 0
Not Completed | 99 | 40
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 17 | 6
Not completed — Study terminated by sponsor | 57 | 24
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Site is closing, site decided to early terminate participant | 1 | 0
Not completed — Missing | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed | Total
Number analyzed (Participants) | 99 | 40 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (15.70) | 41.8 (14.51) | 41.9 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 18 | 65
  Male | 52 | 22 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 23
  Not Hispanic or Latino | 75 | 29 | 104
  Unknown or Not Reported | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 3 | 13
  White | 75 | 34 | 109
  Other | 1 | 1 | 2
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Achieving Clinical Response Measured by Modified Mayo Score for Cohort 1 at Week 12
Description: Clinical response is defined as meeting all of the following improvements from baseline in the Modified Mayo Score:
  * Decrease from baseline ≥ 2 points,
  * Decrease from baseline ≥ 35%,
  * Decrease from baseline in the Rectal Bleeding (RB) subscore ≥ 1 point or absolute RB subscore ≤ 1
  The Modified Mayo Score is a tool that helps doctors measure how active ulcerative colitis is. It combines three components:
  * Stool Frequency (SF): scored 0-3 (higher score = more frequent stools),
  * Rectal Bleeding (RB): scored 0-3 (higher score = more bleeding),
  * Endoscopic Subscore (ES): scored 0-3 (higher score = more severe inflammation seen during endoscopy).
  The total score ranges from 0 to 9, with higher scores meaning more severe disease activity and lower scores meaning less disease activity and better clinical condition.
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 76
  Observed Cases | 65.8 [54.0 to 76.3]
  Non Responder Imputation | 50.5 [40.3 to 60.7]

2. Primary Outcome: Percent of Participants Achieving Clinical Response Measured by Modified Mayo Score for Cohort 2 at Week 26
Description: as for outcome 1
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 25
Percent of Participants | 88.0 [68.8 to 97.5]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any new medical problem or worsening of a preexisting condition in a study participant who receives the study treatment. It does not have to be caused by the treatment. An AE can be any unfavorable and unintended sign (such as an abnormal lab finding), symptom, or disease that happens around the time the study treatment is used, whether or not it is related to the treatment.
  A Treatment Emergent Adverse Event (TEAE) is an AE that meets any of the following:
  * Starts after the first dose of the study treatment (or within 84 days after stopping it) and was not present before; or
  * Was already present before treatment but gets worse after the first dose (or within 84 days after stopping it); or
  * Has missing onset and end dates, making it unclear whether it occurred outside the treatment-emergent period.
  Participants meeting any of these conditions are counted as having at least one TEAE.
Time Frame: From first dose of study medication through post-medication follow-up visit (Up to approximately 812 days)
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 99 | 40
Participants | 61 | 22

4. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, is a congenital anomaly/birth defect, requires in-patient hospitalization or causes prolongation of existing hospitalization, or results in persistent/significant disability/incapacity.
  Treatment Emergent Serious Adverse Event (TE SAE) is a SAE that meets any of the following:
  * Starts after the first dose of the study treatment (or within 84 days after stopping it) and was not present before; or
  * Was already present before treatment but gets worse after the first dose (or within 84 days after stopping it); or
  * Has missing onset and end dates, making it unclear whether it occurred outside the treatment-emergent period.
  Participants meeting any of these conditions are counted as having at least one TESAE.
Time Frame: From first dose of study medication through post-medication follow-up visit (Up to approximately 812 days)
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 99 | 40
Participants | 7 | 4

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event of Interest
Description: This endpoint reports the number of participants who experienced Adverse Events of Interest (AEIs) during the study. AEIs include bradycardia, heart conduction abnormalities (second-degree and higher atrioventricular block), macular edema, malignancy, serious or opportunistic infection, pulmonary effects, hepatic effects, posterior reversible encephalopathy syndrome, progressive multifocal leukoencephalopathy (PML), and events associated with orthostatic hypotension (e.g., dizziness, lightheadedness, syncope, seizure). The Sponsor may request additional information for nonserious AEIs.
  A Treatment Emergent AEI is an AEI that starts after the first dose (or within 84 days after stopping), worsens relative to baseline in this period (or within 84 days after stopping), or has missing dates making the timing unclear.
  Participants meeting any of these conditions are counted as having at least one AEI.
Time Frame: From first dose of study medication through post-medication follow-up visit (Up to approximately 812 days)
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 99 | 40
Participants | 7 | 4

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events Leading to Discontinuation
Description: This endpoint measures the number of participants who experienced Treatment Emergent Adverse Events (TEAEs) that resulted in discontinuation of study treatment.
  An Adverse Event (AE) is any new medical problem or worsening of a preexisting condition in a study participant who receives the study treatment. It does not have to be caused by the treatment. An AE can be any unfavorable and unintended sign (such as an abnormal lab finding), symptom, or disease that happens around the time the study treatment is used, whether or not it is related to the treatment.
  A TEAE is an AE that: starts after the first dose (or within 84 days after stopping) and was not present before; or was preexisting but worsens after the first dose (or within 84 days after stopping); or has missing dates that prevent determining whether it occurred outside the treatment emergent period.
Time Frame: From first dose of study medication through post-medication follow-up visit (Up to approximately 812 days)
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 99 | 40
Participants | 5 | 3

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Assessments
Description: Number of participants experiencing clinically significant abnormalities in laboratory testing including hematology, chemistry and urinalysis.
Time Frame: From first dose of study medication through end of study (Up to approximately 728 days)
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 99 | 40
Participants | 0 | 0

8. Secondary Outcome: Percent of Participants Achieving Clinical Remission by Partial Mayo Score at Week 52 and 104
Description: Clinical remission is defined as a Partial Mayo Score of ≤ 2.5.
  The Partial Mayo Score is a tool that helps doctors measure how active ulcerative colitis is without using endoscopy. It combines three components:
  * Stool Frequency (SF) subscore: range 0-3 (higher score = more frequent stools)
  * Rectal Bleeding (RB) subscore: range 0-3 (higher score = more bleeding)
  * Physician's Global Assessment (PGA): range 0-3 (higher score = worse overall condition based on physician's judgment)
  The total score ranges from 0 to 9, with lower scores meaning fewer symptoms and better disease control, and higher scores meaning more severe disease activity.
  A score of 2.5 or below suggests the disease is in remission.
Time Frame: At week 52 and week 104
Population: Treated participants with observed cases
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 15 | 9
Percent of Participants
  Week 52 - Observed Cases | 80.0 [51.9 to 95.7] | 88.9 [51.8 to 99.7]
  Week 104 - Observed Cases: number analyzed (Participants) | 1 | 2
  Week 104 - Observed Cases | 100.0 [2.5 to 100.0] | 50.0 [1.3 to 98.7]

9. Secondary Outcome: Percent of Participants Achieving Corticosteroid-free Clinical Remission by Partial Mayo Score at Week 52 and 104
Description: Corticosteroid-free Clinical Remission (Partial Mayo Score) is defined as:
  * Meeting the criteria for clinical remission by Partial Mayo Score <=2.5, and
  * No use of oral systemic corticosteroids in the prior 90 days.
  The Partial Mayo Score is a tool that helps doctors measure ulcerative colitis activity without endoscopy. It combines three components:
  * Stool Frequency (SF) subscore: range 0-3 (higher score = more frequent stools)
  * Rectal Bleeding (RB) subscore: range 0-3 (higher score = more bleeding)
  * Physician's Global Assessment (PGA): range 0-3 (higher score = worse overall condition based on physician's judgment)
  The total score ranges from 0 to 9, with lower scores meaning fewer symptoms and better disease control, and higher scores meaning more severe disease activity
Time Frame: At week 52 and week 104
Population: Treated participants with observed cases
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 15 | 9
Percent of Participants
  Week 52 - Observed Cases | 80.0 [51.9 to 95.7] | 77.8 [40.0 to 97.2]
  Week 104 - Observed Cases: number analyzed (Participants) | 1 | 2
  Week 104 - Observed Cases | 100.0 [2.5 to 100.0] | 50.0 [1.3 to 98.7]

10. Secondary Outcome: Percent of Participants Achieving Clinical Response by Partial Mayo Score at Week 52 and 104
Description: Clinical Response by Partial Mayo Score is defined as:
  * Decrease in partial Mayo score ⩾ 2 points and ⩾ 30% from baseline, and
  * Decrease in rectal bleeding subscore > 1 point or absolute rectal bleeding score < 1 This represents a marked improvement in disease activity.
  The Partial Mayo Score is a tool that helps doctors measure ulcerative colitis activity without endoscopy. It combines three components:
  * Stool Frequency (SF) subscore: range 0-3 (higher score = more frequent stools)
  * Rectal Bleeding (RB) subscore: range 0-3 (higher score = more bleeding)
  * Physician's Global Assessment (PGA): range 0-3 (higher score = worse overall condition based on physician's judgment)
  The total score ranges from 0 to 9, with lower scores meaning fewer symptoms and better disease control, and higher scores meaning more severe disease activity.
Time Frame: At week 52 and week 104
Population: Treated participants with observed cases
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 15 | 9
Percent of Participants
  Week 52 - Observed Cases | 93.33 [68.1 to 99.8] | 100.0 [66.4 to 100.0]
  Week 104 - Observed Cases: number analyzed (Participants) | 1 | 2
  Week 104 - Observed Cases | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0]

11. Secondary Outcome: Percent of Participants Achieving Clinical Remission Measured by Modified Mayo Score for Cohort 1 at Week 12
Description: Clinical remission by Modified Mayo Score is defined as meeting all of the following criteria:
  * Stool Frequency (SF) subscore ≤ 1, with at least a 1-point decrease from baseline
  * Rectal Bleeding (RB) subscore = 0
  * Endoscopic Subscore (ES) ≤ 1
  The Modified Mayo Score is the sum of the following components (Range: 0-9):
  * SF subscore: range 0-3 (higher score = more frequent stools)
  * RB subscore: range 0-3 (higher score = more bleeding)
  * ES: range 0-3 (higher score = more severe inflammation seen during endoscopy)
  The total score ranges from 0 to 9, with lower scores meaning less disease activity and better clinical condition, and higher scores meaning more severe disease activity.
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 76
  Observed Cases | 27.6 [18.0 to 39.1]
  Non Responder Imputation | 21.2 [13.6 to 30.6]

12. Secondary Outcome: Percent of Participants Achieving Endoscopic Response for Cohort 1 at Week 12
Description: Endoscopic Response is defined as:
  • A decrease from baseline of ≥ 1 point in the Mayo Endoscopic Score (ES).
  Mayo Endoscopic Score: range 0-3
  * Higher ES scores = more severe inflammation and worse mucosal appearance
  * Lower ES scores = less inflammation and better mucosal healing
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 84
  Observed Cases | 51.2 [40.0 to 62.3]
  Non Responder Imputation | 43.4 [33.5 to 53.8]

13. Secondary Outcome: Percent of Participants Achieving Endoscopic Improvement for Cohort 1 at Week 12
Description: Endoscopic Improvement is defined as:
  • Mayo Endoscopic Score (ES) ≤ 1
  Mayo Endoscopic Score (ES): range 0-3
  * Higher ES scores = more severe inflammation and worse mucosal appearance
  * Lower ES scores = less inflammation and better mucosal healing
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 84
  Observed Cases | 42.9 [32.1 to 54.1]
  Non Responder Imputation | 36.4 [26.9 to 46.6]

14. Secondary Outcome: Percent of Participants Achieving Histological Improvement for Cohort 1 at Week 12
Description: Histological Improvement is defined as:
  • Achieving a Geboes score < 3.1
  The Geboes score is a grading system used to assess inflammation in tissue samples under a microscope.
  * Each domain is graded on a scale, and the total score ranges from 0 to 5.4, with higher scores indicating more severe histologic disease activity.
  * Higher Geboes scores = more severe microscopic inflammation
  * Lower Geboes scores = less inflammation and better healing
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 82
  Observed Cases | 45.1 [34.1 to 56.5]
  Non Responder Imputation | 37.4 [27.9 to 47.7]

15. Secondary Outcome: Change in the Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score From Baseline to Week 12 for Cohort 1
Description: IBDQ is a tool to assess patient experience in inflammatory bowel diseases (Ulcerative Colitis [UC] and Crohn's Disease [CD]).
  It includes 32 questions across 4 dimensions:
  * Bowel symptoms (10 items)
  * Systemic symptoms (5 items)
  * Emotional function (12 items)
  * Social function (5 items)
  Scoring: Each question ranges from 1 ("worst") to 7 ("best"). Total score: 32-224, with higher scores indicating better quality of life (QOL).
  An increase from baseline reflects improved health-related quality of life (HRQOL). The IBDQ is used in registrational studies to evaluate bowel symptoms, functional abdominal symptoms, and overall HRQOL.
Time Frame: At baseline and week 12
Population: Treated participants. Pre-specified to be reported for Cohort 1 only.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 85
Score on a scale | 51.2 (42.86)

16. Secondary Outcome: Percent of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Response [Change in Total Score (≥16 Points) From Baseline to Week 12] for Cohort 1
Description: IBDQ is a tool to assess patient experience in inflammatory bowel diseases (Ulcerative Colitis [UC] and Crohn's Disease [CD]).
  It includes 32 questions across 4 dimensions:
  * Bowel symptoms: 10 items
  * Systemic symptoms: 5 items
  * Emotional function: 12 items
  * Social function: 5 items
  Scoring:
  * Each question ranges from 1 ("worst") to 7 ("best").
  * Total score: 32-224, with higher scores indicating better quality of life (QOL).
  A change from baseline in total score of ≥16 points reflect meaningful IBDQ response. The IBDQ is used in registrational studies to evaluate bowel symptoms, functional abdominal symptoms, and overall health-related quality of life (HRQOL).
Time Frame: At baseline and week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 85
  Observed Cases | 81.2 [71.2 to 88.8]
  Non Responder Imputation | 69.7 [59.6 to 78.5]

17. Secondary Outcome: Percent of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission [Total Score (≥170 Points)] for Cohort 1 at Week 12
Description: IBDQ is a tool to assess patient experience in inflammatory bowel diseases (Ulcerative Colitis [UC] and Crohn's Disease [CD]).
  It includes 32 questions across 4 dimensions:
  * Bowel symptoms: 10 items
  * Systemic symptoms: 5 items
  * Emotional function: 12 items
  * Social function: 5 items
  Scoring:
  * Each question ranges from 1 ("worst") to 7 ("best").
  * Total score: 32-224, with higher scores indicating better quality of life (QOL).
  A total score of ≥170 points reflects IBDQ remission, meaning the participant reports very few symptoms and good overall quality of life. The IBDQ is used in registrational studies to evaluate bowel symptoms, functional abdominal symptoms, and overall health-related quality of life (HRQOL).
Time Frame: At week 12
Population: Treated participants with observed cases and non responder imputation. Pre-specified to be reported for Cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naïve
Number analyzed (Participants) | 99
Percent of Participants
  Observed Cases: number analyzed (Participants) | 89
  Observed Cases | 66.3 [55.5 to 76.0]
  Non Responder Imputation | 59.6 [49.3 to 69.3]

18. Secondary Outcome: Percent of Participants Achieving Clinical Remission Measured by Modified Mayo Score for Cohort 2 at Week 26
Description: as for outcome 11
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 25
Percent of Participants | 68.0 [46.5 to 85.1]

19. Secondary Outcome: Percent of Participants Achieving Endoscopic Response for Cohort 2 at Week 26
Description: Endoscopic Response is defined as:
  • A decrease from baseline of ≥ 1 point in the Mayo Endoscopic Sub score (ES).
  This represents the percentage of treated participants who achieved a decrease from baseline of at least 1 point in the Mayo ES, indicating improvement in mucosal appearance during endoscopy.
  Mayo Endoscopic Subscore (ES): range 0-3
  * Higher ES scores = more severe inflammation and worse mucosal appearance
  * Lower ES scores = less inflammation and better mucosal healing
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 76.7 [57.7 to 90.1]

20. Secondary Outcome: Percent of Participants Achieving Endoscopic Improvement for Cohort 2 at Week 26
Description: Endoscopic Improvement is defined as:
  • Mayo Endoscopic Subscore (ES) ≤ 1
  This represents the percentage of treated participants with Mayo ES ≤ 1, indicating mild or no inflammation.
  Mayo Endoscopic Subscore (ES): range 0-3
  * Higher ES scores = more severe inflammation and worse mucosal appearance
  * Lower ES scores = less inflammation and better mucosal healing
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 63.3 [43.9 to 80.1]

21. Secondary Outcome: Percent of Participants Achieving Endoscopic Remission for Cohort 2 at Week 26
Description: Endoscopic Remission is defined as:
  • Mayo Endoscopic Sub score (ES) = 0
  This represents the percentage of treated participants with Mayo ES = 0, indicating complete mucosal healing.
  Mayo Endoscopic Sub score (ES): range 0-3
  * Higher ES scores = more severe inflammation and worse mucosal appearance
  * Lower ES scores = less inflammation and better mucosal healing
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 33.3 [17.3 to 52.8]

22. Secondary Outcome: Percent of Participants Achieving Histological Improvement for Cohort 2 at Week 26
Description: as for outcome 14
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 63.3 [43.9 to 80.1]

23. Secondary Outcome: Percent of Participants Achieving Histological Remission for Cohort 2 at Week 26
Description: Histological Remission is defined as:
  • Achieving a Geboes score < 2
  The Geboes score is a grading system used to assess inflammation in tissue samples under a microscope.
  * Each domain is graded on a scale, and the total score ranges from 0 to 5.4, with higher scores indicating more severe histologic disease activity.
  * Higher Geboes scores = more severe microscopic inflammation
  * Lower Geboes scores = minimal or no inflammation and better healing
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 53.3 [34.3 to 71.7]

24. Secondary Outcome: Change in the Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score From Baseline to Week 26 for Cohort 2
Description: as for outcome 15
Time Frame: At baseline and week 26
Population: Treated participants. Pre-specified to be reported for Cohort 2 only.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 32
Score on a scale | 63.3 (42.81)

25. Secondary Outcome: Percent of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Response [Change in Total Score (≥16 Points) From Baseline to Week 26] for Cohort 2
Description: as for outcome 16
Time Frame: At baseline and week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 32
Percent of Participants | 84.4 [67.2 to 94.7]

26. Secondary Outcome: Percent of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission [Total Score (≥170 Points)] for Cohort 2 at Week 26
Description: IBDQ is a tool to assess patient experience in inflammatory bowel diseases (Ulcerative Colitis [UC] and Crohn's Disease [CD]).
  It includes 32 questions across 4 dimensions:
  * Bowel symptoms: 10 items
  * Systemic symptoms: 5 items
  * Emotional function: 12 items
  * Social function: 5 items
  Scoring:
  * Each question ranges from 1 ("worst") to 7 ("best").
  * Total score: 32-224, with higher scores indicating better quality of life (QOL).
  A total score of ≥170 points reflect IBDQ remission, meaning the participant reports very few symptoms and good overall quality of life. The IBDQ is used in registrational studies to evaluate bowel symptoms, functional abdominal symptoms, and overall health-related quality of life (HRQOL).
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 33
Percent of Participants | 63.6 [45.1 to 79.6]

27. Secondary Outcome: Percent of Participants Achieving Corticosteroid-free Clinical Remission by Modified Mayo Score for Cohort 2 at Week 26
Description: Corticosteroid-free Clinical Remission (modified mayo score) is defined as:
  * Meeting the criteria for clinical remission by Modified Mayo Score [Stool Frequency (SF) subscore ≤ 1, with ≥ 1 point decrease from baseline and; Rectal Bleeding (RB) subscore = 0 and; Endoscopic Subscore (ES) ≤ 1], and
  * No oral systemic steroid use in the prior 90 days.
  The Modified Mayo Score is the sum of the following components (Range: 0-9):
  * Stool Frequency (SF) subscore: range 0-3 (higher score = more frequent stools)
  * Rectal Bleeding (RB) subscore: range 0-3 (higher score = more bleeding)
  * Endoscopic Subscore (ES): range 0-3 (higher score = more severe inflammation seen during endoscopy)
  The total score ranges from 0 to 9, with:
  * Lower scores = less disease activity and better clinical condition
  * Higher scores = more severe disease activity
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 25
Percent of Participants | 68.0 [46.5 to 85.1]

28. Secondary Outcome: Percent of Participants Achieving Histo-endoscopic Mucosal Improvement (HEMI) for Cohort 2 at Week 26
Description: Histo-endoscopic Mucosal Improvement (HEMI) is defined as:
  * Mayo Endoscopic Subscore (ES) ≤ 1, and
  * Geboes score < 3.1
  Mayo Endoscopic Subscore (ES): range 0-3
  * Higher ES scores = more severe visible inflammation and worse mucosal appearance
  * Lower ES scores = less visible inflammation and better mucosal healing
  Geboes Score:
  * Each domain is graded on a scale, and the total score ranges from 0 to 5.4, with higher scores indicating more severe histologic disease activity
  * Higher Geboes scores = more severe microscopic inflammation
  * Lower Geboes scores = less microscopic inflammation and better tissue healing
  Meeting both criteria (ES ≤ 1 and Geboes < 3.1) shows improvement in both endoscopic appearance and microscopic tissue health.
Time Frame: At week 26
Population: Treated participants with observed cases. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2: Ozanimod Advanced Therapy Exposed
Number analyzed (Participants) | 30
Percent of Participants | 60.0 [40.6 to 77.3]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from first dose to study completion (up to approximately 847 days). SAEs and Other AEs were assessed from first dose of study medication through post-medication follow-up visit (Up to approximately 812 days).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Cohort 1: Ozanimod Advanced Therapy Naive: Advanced therapy naïve participants received ozanimod 0.92 mg daily
Arm/Group | Cohort 1: Ozanimod Advanced Therapy Naive | Cohort 2: Ozanimod Advanced Therapy Exposed
All-Cause Mortality (participants affected / at risk) | 1/99 | 0/40
Serious Adverse Events (participants affected / at risk) | 7/99 | 4/40
Other Adverse Events (participants affected / at risk) | 28/99 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ozanimod Advanced Therapy Naive (N=99) | Cohort 2: Ozanimod Advanced Therapy Exposed (N=40)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ozanimod Advanced Therapy Naive (N=99) | Cohort 2: Ozanimod Advanced Therapy Exposed (N=40)
Colitis ulcerative (Gastrointestinal disorders) | 13 | 4
Nasopharyngitis (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 1
Headache (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT05369832/Prot_SAP_000.pdf